CLINICAL TRIAL: NCT05481294
Title: The Effectivity of Transpersonal Supportive Coaching Intervention on Serotonin Level and Quality of Life in People Living With HIV/AIDS (PLWHA)
Brief Title: Supportive Coaching Intervention in PLWHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Muh. Yusuf Tahir (Other)
Responsible Party: Sponsor-Investigator, Muh. Yusuf Tahir, Lecture, Hasanuddin University
Organization: Hasanuddin University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 683/UN4.6.4.5.31./PP36/2021
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: HIV
Keywords: Serotonin; Quality of Life; Supportive Coaching; PLWHA

STUDY DESIGN:
Intervention Model Description: The intervention group was given transpersonal supportive coaching and ARV therapy. Meanwhile, comparison group 1 was given basic support and ARV therapy, and comparison group 2 was only given ARV therapy without any support.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention with Transpersonal Supportive Coaching (Experimental): PLWHA is given coaching using standard operating procedures (SOP) for Transpersonal Supportive Coaching to encourage or guide patients in obtaining support. The necessary tool is a representative room for two people with two chairs.
  Interventions: Other: Transpersonal Supportive Coaching
- Intervention with Standard Support (Active Comparator): PLWHA is given standard support provided by peer support foundations
  Interventions: Other: Standard Support
- No Support (No Intervention): PLWHA is not given any kind of support

INTERVENTIONS:
Other: Transpersonal Supportive Coaching — Coaching is given for four months (two times a month) with a 45-minute duration per coaching by a professional coach
  Arms: Intervention with Transpersonal Supportive Coaching
Other: Standard Support — Standard support is given for four months using a support system provided by Peer Support Foundation
  Arms: Intervention with Standard Support

SUMMARY:
Introduction:

Coaching is a process of self-exploration, thoughts, and feelings followed by actions within the coachee, through the relationship between the coachee and the coach. This process will help discover potencies in oneself as part of psychological and emotional support.

Objective:

To investigate the effectiveness of Transpersonal Supportive Coaching on Serotonin Levels and Quality of Life PLWHA.

Method:

This research was conducted using an intervention mixed-methods design which is the integration of quantitative and qualitative approaches to study designs, data collections, and analyses.

Alternative hypothesis:

1. There is a difference in serotonin levels before and after Transpersonal Supportive Coaching on PLWHA.
2. There is a difference in the quality of life before and after Transpersonal Supportive Coaching on PLWHA

DETAILED DESCRIPTION:
Sampling technique: Purposive sampling

Sample Size :

The estimation of sample size was calculated using the Slovin formula:

n = N / (1 + (N x e²))

n = sample N = population e = margin error (0.05)

n = 100/(1+100 x 0.0025) = 80

The sample will be divided into 3 groups (each group = 26.67 or 27).

Detailed Intervention:

1. Intervention group: A group was given supportive coaching for 4 months with a 45-minute duration per coaching. It was given two times a month and also taking an antiretroviral (ARV) therapy.
2. Control group I: A group was given only basic support for 4 months and taking ARV therapy.
3. Control group II: A group only taking ARV therapy without any support was given.

Statistical analysis:

1. Qualitative analysis using thematic and content analysis with N-Vivo software
2. Quantitative analysis:

   1. Univariate analysis using Mean and Standard deviation and percentage with 95% Confidence interval
   2. Bivariate analysis using Anova or Kruskal Wallis tests.
   3. Multivariate analysis using logistic regression for main effect test and Process version 5.3.5. for mediation test with bootstrapping method
   4. Data will analysis using SPSS version 26

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed with HIV maximum 2 months
* Stadium I, II

Exclusion Criteria:

* Stadium III and IV
* Opportunistic infection

Drop Out (DO) criteria:

* Not participating in Supportive Coaching for consecutive 3 times
* Not taking ARV for 1 week

Ages: 17 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The change in blood serotonin level | The baseline level of serotonin in blood is measured on the first day before intervention (pre-intervention) and then compared after 4-months of intervention (post-intervention)
  Serotonin (5-hydroxytryptamine, 5-HT) is one of the main neurotransmitters in the human brain that could be affected by psychotherapy (i.e., change the serotonin levels). Total serotonin levels in the blood are measured using the Enzyme-linked Immunoassay (ELISA) method with a standard curve range of 70 ng/L-270 ng/L. The change in serotonin level (i.e., mean score) before and after intervention will be statistically assessed.
The change in Quality of life (QoL) of PLWHA | The baseline score of total and each domain of Quality of Life on PLWHA is measured on the first day before intervention (pre-intervention) and then compared after 4-months of intervention (post-intervention).
  Quality of life is defined as individuals' perception of their position in life in the context of the culture and value system in which they live and in relation to their goals, expectations, standards, and concern which measure using the modified World Health Organization's Quality of Life Questionnaire (WHOQOL-BREF) questionnaire in Indonesian version to measure the QoL patients with HIV/AIDS. it is a 31-item instrument consisting of six domains: physical health (4 items), psychological/emotional well-being (5 items), functional/independence (4 items), social (4 items), environmental (8 items) and spiritual satisfaction (4 items). Further, it also contains overall quality of life and general health perception (2 items). Each item's scores range between 1 (very bad) and 5 (very good). A total score and total of each domain at baseline and after the intervention will be statistically assessed. A positive score change indicates good QoL, while a negative indicates worse QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Tahir, PhD (Cand.), Principal Investigator — Hasanudddin University; Firdaus Hamid, PhD, Study Chair — Hasanudddin University; Risna Halim, PhD, Study Chair — Hasanudddin University; Kusrini S. Kadar, PhD, Study Chair — Hasanudddin University
Locations (1):
- Yayasan Kelompok Dukungan Sebaya (Peer Support Group Foundation), Makassar, South Sulawesi, Indonesia

REFERENCES:
- [Background] Ajisegiri WS, Abubakar AA, Gobir AA, Balogun MS, Sabitu K. Palliative care for people living with HIV/AIDS: Factors influencing healthcare workers' knowledge, attitude and practice in public health facilities, Abuja, Nigeria. PLoS One. 2019 Dec 31;14(12):e0207499. doi: 10.1371/journal.pone.0207499. eCollection 2019. PMID 31891577
- [Background] Bradley PJ, Fureder T, Eckel HE. Systemic Therapy, Palliation and Supportive Care of Patients with Hypopharyngeal Cancer. Adv Otorhinolaryngol. 2019;83:148-158. doi: 10.1159/000492359. Epub 2019 Feb 12. PMID 30943508
- [Background] Burgess MJ, Zeuli JD, Kasten MJ. Management of HIV/AIDS in older patients-drug/drug interactions and adherence to antiretroviral therapy. HIV AIDS (Auckl). 2015 Oct 27;7:251-64. doi: 10.2147/HIV.S39655. eCollection 2015. PMID 26604826
- [Background] Bush SH, Tierney S, Lawlor PG. Clinical Assessment and Management of Delirium in the Palliative Care Setting. Drugs. 2017 Oct;77(15):1623-1643. doi: 10.1007/s40265-017-0804-3. PMID 28864877
- [Background] Busolo D, Woodgate R. Palliative care experiences of adult cancer patients from ethnocultural groups: a qualitative systematic review protocol. JBI Database System Rev Implement Rep. 2015 Jan;13(1):99-111. doi: 10.11124/jbisrir-2015-1809. PMID 26447011
- [Background] Collins AB, Parashar S, Hogg RS, Fernando S, Worthington C, McDougall P, Turje RB, McNeil R. Integrated HIV care and service engagement among people living with HIV who use drugs in a setting with a community-wide treatment as prevention initiative: a qualitative study in Vancouver, Canada. J Int AIDS Soc. 2017 Mar 3;20(1):21407. doi: 10.7448/IAS.20.1.21407. PMID 28426185
- [Background] Gomes B, Calanzani N, Curiale V, McCrone P, Higginson IJ. Effectiveness and cost-effectiveness of home palliative care services for adults with advanced illness and their caregivers. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD007760. doi: 10.1002/14651858.CD007760.pub2. PMID 23744578
- [Background] Harding R, Selman L, Powell RA, Namisango E, Downing J, Merriman A, Ali Z, Gikaara N, Gwyther L, Higginson I. Research into palliative care in sub-Saharan Africa. Lancet Oncol. 2013 Apr;14(4):e183-8. doi: 10.1016/S1470-2045(12)70396-0. PMID 23561750
- [Background] Harding R, Simms V, Alexander C, Collins K, Combo E, Memiah P, Patrick G, Sigalla G, Loy G. Can palliative care integrated within HIV outpatient settings improve pain and symptom control in a low-income country? A prospective, longitudinal, controlled intervention evaluation. AIDS Care. 2013;25(7):795-804. doi: 10.1080/09540121.2012.736608. Epub 2012 Oct 31. PMID 23113572
- [Background] Head BA, Cantrell M, Pfeifer M. Mark's journey: a study in medicaid palliative care case management. Prof Case Manag. 2009 Jan-Feb;14(1):39-45. doi: 10.1097/01.PCAMA.0000343146.81635.38. PMID 19092600
- [Background] Hui D. Definition of supportive care: does the semantic matter? Curr Opin Oncol. 2014 Jul;26(4):372-9. doi: 10.1097/CCO.0000000000000086. PMID 24825016
- [Background] Krakauer EL, Ngoc NT, Green K, Van Kham L, Khue LN. Vietnam: integrating palliative care into HIV/AIDS and cancer care. J Pain Symptom Manage. 2007 May;33(5):578-83. doi: 10.1016/j.jpainsymman.2007.02.004. PMID 17482051
- [Background] Kristanti MS, Setiyarini S, Effendy C. Enhancing the quality of life for palliative care cancer patients in Indonesia through family caregivers: a pilot study of basic skills training. BMC Palliat Care. 2017 Jan 17;16(1):4. doi: 10.1186/s12904-016-0178-4. PMID 28095837
- [Background] McNeil R, Dilley LB, Guirguis-Younger M, Hwang SW, Small W. Impact of supervised drug consumption services on access to and engagement with care at a palliative and supportive care facility for people living with HIV/AIDS: a qualitative study. J Int AIDS Soc. 2014 Mar 13;17(1):18855. doi: 10.7448/IAS.17.1.18855. eCollection 2014. PMID 24629844
- [Background] Medeiros RCDSC, Medeiros JA, Silva TALD, Andrade RD, Medeiros DC, Araujo JS, Oliveira AMG, Costa MAA, Dantas PMS. Quality of life, socioeconomic and clinical factors, and physical exercise in persons living with HIV/AIDS. Rev Saude Publica. 2017 Jul 20;51:66. doi: 10.1590/S1518-8787.2017051006266. PMID 28746573
- [Background] Nkhoma K, Seymour J, Arthur A. An Educational Intervention to Reduce Pain and Improve Pain Management for Malawian People Living With HIV/AIDS and Their Family Carers: A Randomized Controlled Trial. J Pain Symptom Manage. 2015 Jul;50(1):80-90.e4. doi: 10.1016/j.jpainsymman.2015.01.011. Epub 2015 Feb 7. PMID 25666517
- [Background] Qiu J, Jiang YF, Li F, Tong QH, Rong H, Cheng R. Effect of combined music and touch intervention on pain response and beta-endorphin and cortisol concentrations in late preterm infants. BMC Pediatr. 2017 Jan 26;17(1):38. doi: 10.1186/s12887-016-0755-y. PMID 28125980
- [Background] Souza PN, Miranda EJ, Cruz R, Forte DN. Palliative care for patients with HIV/AIDS admitted to intensive care units. Rev Bras Ter Intensiva. 2016 Sep;28(3):301-309. doi: 10.5935/0103-507X.20160054. PMID 27737420
- [Background] Svenningsson I, Petersson EL, Udo C, Westman J, Bjorkelund C, Wallin L. Process evaluation of a cluster randomised intervention in Swedish primary care: using care managers in collaborative care to improve care quality for patients with depression. BMC Fam Pract. 2019 Jul 27;20(1):108. doi: 10.1186/s12875-019-0998-4. PMID 31351444